CLINICAL TRIAL: NCT04342130
Title: Brain Effects of Opiate Agonist and Antagonist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Paul Geha, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YaleIRB#1607018141
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): People with low back pain who were given and oral dose of 30 mg morphine.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 30 mg oral tablet

SUMMARY:
This study will look at the short-term effect of morphine on brain response to food.

DETAILED DESCRIPTION:
Chronic low back pain patients and healthy controls will be recruited for this study. Participants' brain will be scanned at baseline and then again on a different day after the administration of an oral dose of 30 mg morphine in an open label design. Participants will receive morphine 60 minutes prior to the start of the second scanning session. The brain scans will include structural scans, functional scans at rest and functional scans during the ingestion of a highly caloric drink.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Patients in pain: suffering from persistent pain more days than not, 3/10 in intensity on a numerical rating scale, for at least 6 weeks or more.

Exclusion Criteria:

* Any DSM diagnosis
* diabetes
* food allergies
* lactose intolerance
* participants seeking to quit smoking or to lose weight
* participants on any psychotropic medication including opiate based analgesics (e.g. oxycodone, methadone, suboxone)
* pregnant or nursing women
* pacemaker or other implanted electrical devices
* Participants with a past history of head trauma or seizures
* Any past history of illegal drug or alcohol misuse
* Participants who cannot undergo an MRI scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Geha, MD, Principal Investigator — Department of Psychiatry in University of Rochester
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data available from this trial will made available to researcher via reasonable request from the PI.
Supporting Information: Study Protocol, SAP
Time Frame: study protocol and analytic code will be available after manuscript publication
Access Criteria: Upon reasonable request from the PI

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 mg Morphine: People with low back pain who were given and oral dose of 30 mg morphine.
  Morphine: 30 mg oral tablet
Period: Overall Study
Arm/Group | 30 mg Morphine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 30 mg Morphine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Subcortical Brain Structure Volume
Description: Magnetic Resonance Imaging (MRI) scanning was performed to collect brain volume measurements in cc. There were 4 different areas of the brain that were analyzed.
Time Frame: baseline to 1 hour
Population: One participant was missing data for this outcome measure.
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | 30 mg Morphine
Number analyzed (Participants) | 9
cubic centimeters
  nucleus accumbens | 0.054 (0.36)
  thalamus | 0.74 (2.8)
  amygdala | 0.27 (0.38)
  hippocampus | 0.48 (1.4)
Statistical Analysis 1: Comparison: 30 mg Morphine; Test type: Other; p > 0.05, t-test, 2 sided

2. Primary Outcome: Change in Brain Response to Highly Caloric Drink
Description: Participants received a highly caloric drink and a tasteless solution during a functional MRI scanning session. A general linear model was used to generate the magnitude of the fit for each type of stimuli and differences between the fits were calculated. A within subject analysis approach was used to calculate the effect of an acute dose of morphine on brain response to the highly caloric drink. Participants contributed beta values that were averaged across subjects and based on the average and standard deviation, the software, FSL, calculated Z = 4.38. This value indicates 4.38 standard deviations away from the mean in a distribution with a mean of zero and standard deviation of 1, which is the definition of the Gaussian curve (Z-distribution). It is scientifically not valid to say there is a higher or lower brain response. A Z-score = 0 means no change from baseline in brain response; a Z-score different from zero indicates a change from baseline after the ingestion of morphine.
Time Frame: baseline to 1 hour
Measure: Number; unit: z-score
Arm/Group | 30 mg Morphine
Number analyzed (Participants) | 10
z-score | 4.38

3. Primary Outcome: Mean Change in Resting Brain Activity in the Nucleus Accumbens
Description: Participants were scanned at rest during a functional MRI session. The resting brain activity was measured as the Power spectral density slow-4 frequency band. Data collected in the frequency range 0 and 0.5 Hertz was analyzed. We examined the power spectral density in the range of 0.027 to 0.073 Hertz. The mean change is expressed as arbitrary units after a Fourier transformation of the data which cancels out the units. The mean change ranges from 0 to 175. The higher the number the more energy within that frequency band.
Time Frame: baseline to 1 hour
Population: Data was missing for one participant for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 30 mg Morphine
Number analyzed (Participants) | 9
units on a scale | 14.5 (10.4)

4. Secondary Outcome: Mean Change in Back Pain Intensity
Description: Pain was rated using a visual analog scale ranging from 0-100 with 100 indicating the worst imaginable pain ever.
Time Frame: baseline to 1 hour
Population: Back pain data was missing for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 30 mg Morphine
Number analyzed (Participants) | 9
units on a scale | 3.6 (1.7)

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | 30 mg Morphine
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 30 mg Morphine (N=10)
Itching (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT04342130/Prot_SAP_001.pdf
  • Informed Consent Form (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT04342130/ICF_000.pdf